CLINICAL TRIAL: NCT07019402
Title: Internet-based Mind-Body Training (iMBT) for Brain Health
Brief Title: Internet-based Mind-Body Training for Brain Health
Acronym: iMBT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024H0401; 1R61AG081982-01A1 (NIH)
Record Dates: First submitted 2025-04-07; First posted 2025-06-13 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Subjective Cognitive Decline
Keywords: mindfulness-based stress reduction; mind-wandering; mind-body training; aging; subjective cognitive decline; lifestyle education; randomized control trial

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Single-blind. Any investigators administering assessments will be blind to participants' group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based Mindfulness-Based Stress Reduction (iMBSR) (Experimental): Participants will access mindfulness exercises using the ScarletCanvas platform and will complete them at their own pace throughout the intervention. The iMBSR protocol is developed to ensure that participants spend 2.5 hrs/week on each of the eight modules. The protocol will have a mix of didactics, experiential practices, social support, and community building. Experiential practices in iMBSR will include body scans, sitting meditations, and mindful movement.
  Interventions: Behavioral: Internet-based Mindfulness-Based Stress Reduction (iMBSR)
- Internet-based Lifestyle Education Group (iLifeEd) (Active Comparator): Participants will access lifestyle education exercises using the ScarletCanvas platform and will complete them at-their own pace throughout the intervention. The iLifeEd protocol is developed to ensure that participants spend 2.5 hrs/week on each of the eight modules. The protocol will have a mix of didactics, experiential practices, social support, and community building. Experiential practices in iLifeEd will include stretching and toning exercises matched in duration to the practices of iMBSR.
  Interventions: Behavioral: Internet-based Lifestyle Education (iLifeEd)

INTERVENTIONS:
Behavioral: Internet-based Mindfulness-Based Stress Reduction (iMBSR) — The iMBSR program is an adaptation of Jon Kabat-Zinn's Mindfulness-Based Stress Reduction (MBSR) to be delivered in an online and asynchronous manner. MBSR was developed by Kabat-Zinn in the 1970s as a method to help individuals manage stress and pain through mindfulness meditation. Mindfulness practice has been linked to numerous benefits such as boosting cognitive control and emotion regulation. MBSR includes practices such as orienting attention to the present moment, often through an object like the breath, nonjudgmental awareness of thoughts and emotions, mindful listening, mindful eating, and body scan meditation.
  Arms: Internet-based Mindfulness-Based Stress Reduction (iMBSR)
Behavioral: Internet-based Lifestyle Education (iLifeEd) — iLifeEd is an online and asynchronous lifestyle education program. Participants will be presented with information and activities about healthy aging topics, including physical activity, sedentary behavior, sleep, stress, nutrition and hydration, social support, and cognitively stimulating activities. Stretching and toning exercises will also be included.
  Arms: Internet-based Lifestyle Education Group (iLifeEd)

SUMMARY:
The goal of this study is to conduct a Stage I pilot study examining the feasibility, acceptability, and preliminary effects of an internet-based, asynchronous mindfulness-based stress reduction program (iMBSR) compared to an internet-based, asynchronous lifestyle education program (iLifeEd), for adults at-risk for Alzheimer's disease (AD). Sixty middle-aged and older adults (aged 50 years or older) with subjective cognitive decline will be randomized to either an 8-week iMBSR program or an 8-week iLifeEd program control group, designed to provide adequate control for placebo effects. Behavioral, neuroimaging, and ecological momentary assessment (EMA) measures of mind-wandering will be administered to determine preliminary effects as a function of engagement in the iMBSR program. AD biomarkers will be examined at pre-training and post-training assessments.

DETAILED DESCRIPTION:
A significant limiting factor in the prognosis of AD is the absence of targeted pharmaceutical or behavioral interventions to arrest or reduce the neurodegeneration resulting from the accumulation of two key proteinopathies once cognitive symptoms are observable. In fact, in AD stage sequencing, the aggregation of Aβ in neural plaques followed by tau accumulation in neurofibrillary tangles, predates the onset of known cognitive symptoms-at times one to two decades before observable changes in cognition. Additionally, midline cortical structures of the DMN are the first sites of AD pathophysiology with activity of the DMN heavily linked with internally directed cognitions. Although these internally directed cognitions are adaptive, the ongoing nature of these spontaneous cognitions has a downstream negative impact for overall cognition, psychological well-being, and potentially, is also linked with AD pathophysiology. Mindfulness training, with its cultivation of present moment awareness, has shown promising support for its potential to reduce mind-wandering and strengthen the neural circuitry supporting sustained attention. More recently, there has also been support for mindfulness to be positively associated with lower levels of Aβ and tau pathology. Thus, the primary goal of this study is to evaluate the feasibility, acceptability, and preliminary effects of an internet-based mindfulness training program on mind-wandering, neural connectivity of the DMN, and plasma-based biomarkers of Aβ and tau pathology, which has the potential to make a significant contribution to the prevention of AD-related cognitive decline. The main hypothesis is that the iMBSR program will be feasible and acceptable and improve neural, behavioral, and EMA measures of mind-wandering and slow the accumulation of AD biomarkers. Feasibility will be defined through evaluation of recruitment, retention, and drop-out rates. Acceptability will be defined by assessing prospective acceptability, participant attendance, and program satisfaction. The investigators hypothesize that iMBSR and iLifeEd will be feasible and acceptable for adults with subjective cognitive decline, and that participants in the iMBSR group will also report lower levels of subjective cognitive decline. The investigators additionally hypothesize that iMBSR training will result in a reduction of mind-wandering thoughts and reaction time coefficient of variation (RT_CV) immediately following training. The investigators also hypothesize that network strength in the default mode network (DMN) will increase following training in the iMBSR protocol compared with the iLifeEd training. For plasma markers of amyloid and tau pathology, the investigators hypothesize that there will be a lower rate of accumulation in amyloid and tau pathology in the iMBSR group compared with the iLifeEd group.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years or greater
* Capable of attending screening and assessment sessions and the internet-based intervention modules
* Fluent English speaker
* Corrected (near and far) visual acuity of 20/40 or better
* Adequate hearing for experimental purposes
* Absence of diagnosed terminal illness
* Absence of diagnosed neurological disorders
* No history of psychotic disorder or substance abuse disorder diagnosed by a psychologist or psychiatrist
* Absence of medication use that significantly alters brain activity
* No history of diagnosed learning disability that would interfere with the completion of the cognitive tasks
* Report elevated scores on the self-report Everyday Cognition (E-Cog)-39 subjective cognitive decline with normatively intact performance on cognitive testing (as determined by the neuropsychological battery)
* No evidence of mild cognitive impairment or dementia as assessed by the neuropsychological measures from the National Alzheimer's Coordinating Center (NACC) Uniform Data Set OR inadequate self-reported performance of instrumental activities of daily living
* Ability to engage in light stretching/movement-based activities with or without assistive devices
* Absence of any MRI contraindications
* Not pregnant and not attempting to become pregnant
* Absence of self-reported claustrophobia
* No regular practice of meditation or yoga (defined as once or more per week) AND No previous participation in a structured mindfulness class (e.g., Mindfulness-Based Stress Reduction, intensive meditation retreat)
* Access to internet and at-home computer with a working microphone and video
* Not enrolled in other RCTs examining the efficacy of exercise training, cognitive rehabilitation, stress management, progressive muscle relaxation or other health-based rehabilitation

Exclusion Criteria:

* Aged less than 50 years
* Any physical or pragmatic limitation that prohibits attendance of screening or assessment sessions, or intervention engagement
* No fluency in English
* Corrected (near or far) visual acuity worse than 20/40
* Self-reported hearing impairment that would affect ability to hear the experimenter
* Diagnosis of terminal illness
* Presence of diagnosed neurological disorders such as: Alzheimer's disease, Vascular Dementia, Parkinson's disease, Multiple Sclerosis, Traumatic Brain Injury, Fronto-Temporal Lobar Degeneration, Lewy Body Disease
* History of psychotic disorder or substance abuse disorder diagnosed by a psychologist or psychiatrist
* Medication use that significantly alters brain activity
* History of diagnosed learning disability that would interfere with the completion of the cognitive tasks
* Does not report subjective cognitive decline AND/ OR does not perform in the normatively intact range on neuropsychological testing
* Evidence of mild cognitive impairment (MCI) or dementia OR inadequate self-reported performance of instrumental activities of daily living
* Any physical limitation or pragmatic limitation that prohibits attendance at assessment sessions and intervention modules with or without assistive devices
* Presence of MRI contraindications as assessed through the MRI screening form.
* Pregnant or attempting to become pregnant
* Self-reported claustrophobia
* Any regular practice of meditation or yoga (defined as once or more per week) OR Previous participation in a structured mindfulness class (e.g., Mindfulness-Based Stress Reduction, intensive meditation retreat)
* No access to internet or at-home computer with a working microphone and video
* Current enrollment in other RCTs examining the efficacy of exercise training, cognitive rehabilitation, stress management, progressive muscle relaxation or other health-based rehabilitation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of intervention: Recruitment | 12 months
  Feasibility will be determined by evaluating the recruitment of study participants. High feasibility will be defined as the successful recruitment of 60 participants over one year.
Feasibility of intervention: Retention rate | 8 weeks
  Feasibility will be determined by evaluating retention of participants in the study.
Feasibility of intervention: attrition rate | 8 weeks
  High feasibility will be defined as an attrition rate of enrolled participants of no greater than 25%.
Acceptability of intervention | 8 weeks
  Prospective acceptability will be assessed using the Acceptability of Intervention Measure (AIM). High acceptability will be defined as an average score greater than 3 (on a 1-5, completely agree-completely disagree scale).
Program satisfaction | 8 weeks
  Program satisfaction will be measured by our custom Post-Intervention Acceptability Questionnaire which focuses on program enjoyment and satisfaction and potential barriers. High program satisfaction will be defined as an average score greater than 5 (on a 0-10, not at all-extremely scale) for items focused on satisfaction.
Participant attendance | 8 weeks
  Participant attendance will be determined by data on module completion on the class platform ScarletCanvas. High participation will be defined as at least 50% of participants successfully completing 6 or more modules.
Changes in subjective cognitive decline | Baseline, 8 weeks
  Participants will be administered the self-report Everyday Cognition Questionnaire (ECog) at pre-intervention and post-intervention. Significant changes in subjective reports of cognitive decline will also be considered as evidence for feasibility of the intervention.
Plasma-based Alzheimer's disease (AD) biomarkers | Baseline, 8 weeks
  Plasma markers of amyloid and tau pathology will be assayed at pre-intervention and post-intervention.

SECONDARY OUTCOMES:
Default mode network (DMN) strength | Baseline, 8 weeks
  Network strength in the DMN during the Gradual-onset Continuous Performance Task (GradCPT) will be computed from the MRI scans at pre-intervention and post-intervention.
Behavioral measure of Mind-wandering | Baseline, 8 weeks
  The primary measure of mind-wandering will be the reaction time coefficient of variation (RT_CV), which will be obtained by computing the trial to trial fluctuations in participant reaction time during the Go/No-Go task at pre-intervention and post-intervention.
Self-report measures of Mind-wandering | Baseline, 8 weeks
  The primary measure of self-reported mind-wandering will be the self-report endorsement of mind-wandering during daily life collected during ecological momentary assessment (EMA) at pre-intervention and post-intervention.

OTHER OUTCOMES:
Self-report stress | Baseline, 8 weeks
  The Perceived Stress Scale (PSS) will be administered pre-intervention and post-intervention to measure self-report perceptions of stress. The measure has 10 items measured on a 5-point scale. Total score is obtained by summing individual item scores, with a higher score indicating greater stress.
Self-report motivation to change life style and health behaviors for dementia risk reduction | Baseline, 8 weeks
  The Motivation to Change Lifestyle and Health Behaviors for Dementia Risk Reduction Scale (MCLHB-DRR) will be administered pre-intervention and post-intervention to assess self-report motivation to change life style and health behaviors for dementia risk reduction. The measure has 27 items measured on a 5-point scale. Total score is obtained by summing individual item scores, with a higher score indicating greater motivation.
Self-report quality of life | Baseline, 8 weeks
  The World Health Organization Quality of Life abbreviated scale (WHOQOL-BREF) will be administered pre-intervention and post-intervention to assess self-reported quality of life. The measure has 26 items scored on a 5-point scale. Total score is obtained by summing individual item scores, with a higher score indicating greater quality of life.
Self-report anxiety | Baseline, 8 weeks
  The Beck Anxiety Inventory (BAI) will be administered pre-intervention and post-intervention to assess self-report anxiety. The measure has 21 items measured on a 4-point scale. Total score is obtained by summing individual item scores, with a higher score indicating greater anxiety.
Self-report worry | Baseline, 8 weeks
  The Penn State Worry Questionnaire (PSWQ) will be administered pre-intervention and post-intervention to assess self-report worry. The measure has 16 items measured on a 5-point scale. Total score is obtained by summing individual item scores (with 5 items reverse-scored), with a higher score indicating greater worry.
Self-report discrimination | Baseline, 8 weeks
  The Everyday Discrimination Scale (EDS) will be administered pre-intervention and post-intervention to assess self-report accounts of everyday discrimination. The measure has 9 required items scored on a 6-point scale. Total score is obtained by summing individual item scores, with a higher score indicating greater discrimination.
Self-report depression | Baseline, 8 weeks
  The Center for Epidemiological Studies-Depression Scale (CES-D) will be administered pre-intervention and post-intervention to assess self-report depression. The measure has 20 items scored on a 4-point scale. Total score is obtained by summing individual item scores (with 4 items reverse-scored), with a higher score indicating greater depression.
Intra-individual variability in EMA-based cognitive functioning | Baseline, 8 weeks
  Participants will complete ecological momentary assessment of cognitive functioning before and immediately after the intervention. We will compute intraindividual variability in cognitive performance to examine the effect of the intervention.
Hippocampal Volume | Baseline, 8 weeks
  Hippocampal volume will be computed using a high-resolution MRI scan. Multi-spectral analyses, employing the Automatic Segmentation of Hippocampal Subfields, will be conducted to quantify volumetric changes in the hippocampal subfields.

CONTACTS AND LOCATIONS:
Overall Officials: Ruchika S Prakash, PhD, Principal Investigator — Ohio State University
Locations (1):
- Department of Psychology, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Warburton DE, Jamnik VK, Bredin SS, McKenzie DC, Stone J, Shephard RJ, Gledhill N. Evidence-based risk assessment and recommendations for physical activity clearance: an introduction. Appl Physiol Nutr Metab. 2011 Jul;36 Suppl 1:S1-2. doi: 10.1139/h11-060. PMID 21800937
- [Background] Bondi MW, Edmonds EC, Jak AJ, Clark LR, Delano-Wood L, McDonald CR, Nation DA, Libon DJ, Au R, Galasko D, Salmon DP. Neuropsychological criteria for mild cognitive impairment improves diagnostic precision, biomarker associations, and progression rates. J Alzheimers Dis. 2014;42(1):275-89. doi: 10.3233/JAD-140276. PMID 24844687
- [Background] Jack CR Jr, Knopman DS, Jagust WJ, Petersen RC, Weiner MW, Aisen PS, Shaw LM, Vemuri P, Wiste HJ, Weigand SD, Lesnick TG, Pankratz VS, Donohue MC, Trojanowski JQ. Tracking pathophysiological processes in Alzheimer's disease: an updated hypothetical model of dynamic biomarkers. Lancet Neurol. 2013 Feb;12(2):207-16. doi: 10.1016/S1474-4422(12)70291-0. PMID 23332364
- [Background] Sperling RA, Aisen PS, Beckett LA, Bennett DA, Craft S, Fagan AM, Iwatsubo T, Jack CR Jr, Kaye J, Montine TJ, Park DC, Reiman EM, Rowe CC, Siemers E, Stern Y, Yaffe K, Carrillo MC, Thies B, Morrison-Bogorad M, Wagster MV, Phelps CH. Toward defining the preclinical stages of Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):280-92. doi: 10.1016/j.jalz.2011.03.003. Epub 2011 Apr 21. PMID 21514248
- [Background] Strikwerda-Brown C, Ozlen H, Pichet Binette A, Chapleau M, Marchant NL, Breitner JCS, Villeneuve S. Trait Mindfulness Is Associated With Less Amyloid, Tau, and Cognitive Decline in Individuals at Risk for Alzheimer's Disease. Biol Psychiatry Glob Open Sci. 2022 Jan 17;3(1):130-138. doi: 10.1016/j.bpsgos.2022.01.001. eCollection 2023 Jan. PMID 36712573
- [Background] Tomaszewski Farias S, Mungas D, Harvey DJ, Simmons A, Reed BR, Decarli C. The measurement of everyday cognition: development and validation of a short form of the Everyday Cognition scales. Alzheimers Dement. 2011 Nov;7(6):593-601. doi: 10.1016/j.jalz.2011.02.007. PMID 22055976
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Sperling R, Mormino E, Johnson K. The evolution of preclinical Alzheimer's disease: implications for prevention trials. Neuron. 2014 Nov 5;84(3):608-22. doi: 10.1016/j.neuron.2014.10.038. Epub 2014 Nov 5. PMID 25442939
- [Background] Yiannopoulou KG, Papageorgiou SG. Current and Future Treatments in Alzheimer Disease: An Update. J Cent Nerv Syst Dis. 2020 Feb 29;12:1179573520907397. doi: 10.1177/1179573520907397. eCollection 2020. PMID 32165850
- [Background] Weintraub S, Besser L, Dodge HH, Teylan M, Ferris S, Goldstein FC, Giordani B, Kramer J, Loewenstein D, Marson D, Mungas D, Salmon D, Welsh-Bohmer K, Zhou XH, Shirk SD, Atri A, Kukull WA, Phelps C, Morris JC. Version 3 of the Alzheimer Disease Centers' Neuropsychological Test Battery in the Uniform Data Set (UDS). Alzheimer Dis Assoc Disord. 2018 Jan-Mar;32(1):10-17. doi: 10.1097/WAD.0000000000000223. PMID 29240561
- [Background] Schultz AP, Chhatwal JP, Huijbers W, Hedden T, van Dijk KR, McLaren DG, Ward AM, Wigman S, Sperling RA. Template based rotation: a method for functional connectivity analysis with a priori templates. Neuroimage. 2014 Nov 15;102 Pt 2(0 2):620-36. doi: 10.1016/j.neuroimage.2014.08.022. Epub 2014 Aug 21. PMID 25150630
- [Background] Martinon LM, Smallwood J, McGann D, Hamilton C, Riby LM. The disentanglement of the neural and experiential complexity of self-generated thoughts: A users guide to combining experience sampling with neuroimaging data. Neuroimage. 2019 May 15;192:15-25. doi: 10.1016/j.neuroimage.2019.02.034. Epub 2019 Feb 22. PMID 30802513
- [Background] Lutz A, Jha AP, Dunne JD, Saron CD. Investigating the phenomenological matrix of mindfulness-related practices from a neurocognitive perspective. Am Psychol. 2015 Oct;70(7):632-58. doi: 10.1037/a0039585. PMID 26436313
- [Background] Jak AJ, Bondi MW, Delano-Wood L, Wierenga C, Corey-Bloom J, Salmon DP, Delis DC. Quantification of five neuropsychological approaches to defining mild cognitive impairment. Am J Geriatr Psychiatry. 2009 May;17(5):368-75. doi: 10.1097/JGP.0b013e31819431d5. PMID 19390294
- [Background] Gauthier S, Albert M, Fox N, Goedert M, Kivipelto M, Mestre-Ferrandiz J, Middleton LT. Why has therapy development for dementia failed in the last two decades? Alzheimers Dement. 2016 Jan;12(1):60-4. doi: 10.1016/j.jalz.2015.12.003. Epub 2015 Dec 19. PMID 26710325
- [Background] Farias ST, Mungas D, Reed BR, Cahn-Weiner D, Jagust W, Baynes K, Decarli C. The measurement of everyday cognition (ECog): scale development and psychometric properties. Neuropsychology. 2008 Jul;22(4):531-44. doi: 10.1037/0894-4105.22.4.531. PMID 18590364
- [Background] Boot WR, Charness N, Czaja SJ, Sharit J, Rogers WA, Fisk AD, Mitzner T, Lee CC, Nair S. Computer proficiency questionnaire: assessing low and high computer proficient seniors. Gerontologist. 2015 Jun;55(3):404-11. doi: 10.1093/geront/gnt117. Epub 2013 Oct 9. PMID 24107443